CLINICAL TRIAL: NCT00784264
Title: A Study on Intima Media Thickness (IMT) in Middle-aged Subjects
Acronym: IMT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Karen Yuen, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CHK-DUM-2008/1
Record Dates: First submitted 2008-10-22; First posted 2008-11-03 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Atherosclerosis
Keywords: Asymptomatic atherosclerosis; Intima media thickness (IMT); central obesity; cardiovascular disease
MeSH Terms: conditions — Atherosclerosis; Obesity, Abdominal; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to measure the thickness of artery walls in the neck (intima media thickness IMT) by ultrasound examination in middle-aged subjects with central obesity. The purpose of this study is to obtain local data how common asymptomatic atherosclerosis is, and to investigate the association between Cardiovascular Disease risk factors and intima media thickness (IMT) in the Hong Kong population. Results from this study may enhance the public awareness of asymptomatic atherosclerosis and understand its role in the development of Cardiovascular Disease in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 55 years or above.
* Waist circumference: male more than 90 cm; female more than 80 cm.

Exclusion Criteria:

* Any known chronic diseases requiring long-term medication such as hypertension, diabetes and hyperlipidemia.
* Presence of known cardiovascular diseases including cerebro-vascular disease, coronary heart disease and peripheral artery disease.
* Presence of any active major diseases that may interfere the physical conditions and body weight of subjects during the study period, which include malignancy, infection, renal or liver function impairment, recent major surgery (within 3 months).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: aged 55 or above with central obesity, male more than 90 cm; female more than 80 cm
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-10; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To investigate the prevalence of asymptomatic atherosclerosis by measurement of intima media thickness (IMT) in middle-aged subjects with central obesity in Hong Kong, | during the one single study visit

SECONDARY OUTCOMES:
To examine the association between IMT value and cardiovascular disease (CVD) risk factors, and blood lipid and glucose profiles in middle-aged centrally obese subjects in Hong Kong. | During the one single study visit
IMT results to be compared with what being reported in the recent literature on normal Chinese population. | During the one single study visit

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yuen, Study Director — AstraZeneca Hong Kong Ltd; Chun chung Chow, MD, Principal Investigator — Prince of Wales Hospital, Shatin, Hong Kong
Locations (1):
- Research Site, Hong Kong, Hong Kong